CLINICAL TRIAL: NCT03539887
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of the Rapid Antisuicidal Effects of Intranasal Ketamine in Comorbid Depression and Alcohol Abuse
Brief Title: Trial of the Rapid Antisuicidal Effects of Intranasal Ketamine in Comorbid Depression and Alcohol Abuse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rodrigo Machado-Vieira, MD, PhD, MSc, Professor of Psychiatry, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-17-0903
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Suicidal Ideation; Depression; Alcohol Abuse
Keywords: Ketamine; Depression; Suicidal Ideation; Alcohol Abuse
MeSH Terms: conditions — Suicidal Ideation; Depression; Alcoholism

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal ketamine (Experimental): Intranasal ketamine
  Interventions: Drug: Intranasal ketamine
- Placebo (Placebo Comparator): non-active placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal ketamine — Intranasal ketamine will be prepared as 100mg/ml ketamine in 0.9% saline. An mucosal atomization device will be used to provide 5 intranasal applications of solution (volume 100 μl), separated by 3 minutes, over a total of 15 minutes. Each of five ketamine applications will provide 10 mg of study drug, for a total of 50mg. The dose to be used (0.5-1mg/Kg) is 6 to 18 times lower than the sedation dose (6-9mg/Kg).
  Arms: Intranasal ketamine
Drug: Placebo — Saline alone. An mucosal atomization device will be used to provide 5 intranasal applications of saline (volume 100 μl), separated by 3 minutes, over a total of 15 minutes.
  Arms: Placebo

SUMMARY:
This project aims to evaluate the potential rapid and sustained antisuicidal and antidepressant effects of a single intranasal dose of ketamine in inpatients during a mood episode in Major Depressive Disorder (MDD) or Bipolar Disorder (BD) with or without comorbid recent abuse of alcohol.

DETAILED DESCRIPTION:
Clinicians have a limited ability to predict imminent suicidal behavior and efficacious treatments are not available to treat suicidal patients. Thus, Rapid-acting treatments for suicidal individuals are truly needed. This project aims to evaluate the potential rapid and sustained antisuicidal and antidepressant effects of a single intranasal dose of ketamine in inpatients during a mood episode (in Major Depressive Disorder, MDD or Bipolar Disorder, BD) with or without comorbid recent abuse of alcohol. These results will elucidate the antisuicidal effects of ketamine using the intranasal route along with the identification of associated mediators or moderators; this approach has the potential for enormous public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary admission to Harris County Psychiatry Center
* Able to provide written informed consent
* Current suicidal ideation and depressive symptoms and Diagnostic and Statistical Manual of Mental Disorders -IV- Text Revision(DSM-IV-TR) depressive episode (also MADRS greater than or equal to 12) and Young Mania Rating Scale (YMRS) score lower than 8
* DSM-IV-TR criteria for current alcohol abuse (but not intoxicated/withdrawal, abstinent from drinking for > 5 days prior to admission).
* Lifetime history of suicide attempt (patient)
* Not taking any medication in the last 24hs.
* Scale for Suicide Ideation (SSI) score over 4 (first five items) and Columbia scale (C-SSRS) score 4 or 5

Exclusion Criteria:

* Unstable medical condition or medical problem with known central nervous system (CNS) effects, e.g. uncontrolled hypertension systolic blood pressure (SBP) ≥170 and/or diastolic blood pressure (DBP) ≥100) or recent history (6 months) of alcohol-withdrawal seizures or significant abnormal laboratory tests (liver function test (LFT) 3 times higher than normal).
* Prior diagnosis of a DSM-IV-TR psychotic spectrum disorder, psychotic symptoms, or personality disorder.
* Currently under the acute effects of an illicit substance.
* Pregnant or nursing women.
* Subjects with a history of DSM-IV drug dependency or abuse (except for caffeine or nicotine dependence) within the preceding 3 months

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Machado-Vieira, MD, PhD, MSc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Jones GH, Vecera CM, Ruiz AC, Wu HE, McInturff SI, Orejarena MJ, Smith KA, Soares JC, Zarate CA, Lane SD, Machado-Vieira R. A Randomized, Double-Blind, Placebo-Controlled Pilot Trial of the Acute Antisuicidal and Antidepressant Effects of Intranasal (R,S)-Ketamine in Severe Unipolar and Bipolar Depression With and Without Comorbid Alcohol Use Disorder. J Clin Psychiatry. 2024 Apr 24;85(2):23m14974. doi: 10.4088/JCP.23m14974. PMID 38696221
- See also: Department of Psychiatry, Dr Rodrigo Machado-Vieira — https://med.uth.edu/psychiatry/faculty/rodrigo-machado-vieira-m-d-ph-d-m-sc/
- See also: Experimental Therapeutics and Molecular Pathophysiology, UTHealth, Houston, Texas — https://med.uth.edu/psychiatry/research/programs/experimental-therapeutics-molecular-pathophysiology-program/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants who were enrolled were not randomized and did not start the study.
Period: Overall Study
Arm/Group | Intranasal Ketamine | Placebo
Started | 17 | 11
Completed | 17 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Ketamine | Placebo | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (9) | 38.5 (13.8) | 38.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Suicidal Ideation as Assessed by the Scale for Suicide Ideation (SSI)
Description: The scale contains 19 items rated on a scale from 0 to 2, allowing score range from 0 to 38, score over 4 (first five items) will be considered inclusion criteria. Higher values indicate worsening or presence of suicidal ideation.
Time Frame: 24 hours
Population: Data for this outcome measure were not collected for 1 participant in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Ketamine | Placebo
Number analyzed (Participants) | 17 | 10
score on a scale | 10.8 (8.08) | 12.3 (7.83)

2. Secondary Outcome: Depression as Assessed by the Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: It has ten items, each item yields a score of 0 to 6. Hence the overall score ranges from 0 to 60. Higher scores indicate more severe depression.
Time Frame: 24 hours
Population: Data for this outcome measure were not collected for 1 participant in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Ketamine | Placebo
Number analyzed (Participants) | 17 | 10
score on a scale | 16.8 (13.7) | 22.5 (17.7)

3. Secondary Outcome: Snaith-Hamilton Pleasure Scale
Description: The Snaith-Hamilton Pleasure Scale (SHAPS) is an assessment of anhedonia, which is the inability to experience pleasure. The SHAPS has 14 items. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. A response of "strongly disagree" or "disagree" equals one point, and a response of "strongly agree" or "agree" equals 0 points. Thus, the final score ranges from 0 to 14. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more.
Time Frame: 24 hours
Population: Data for this outcome measure were not collected for 1 participant in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Ketamine | Placebo
Number analyzed (Participants) | 17 | 10
score on a scale | 4.12 (4.81) | 5.00 (4.29)

4. Secondary Outcome: Alcohol Urge Questionnaire (AUQ)
Description: Alcohol Urge Questionnaire (AUQ) is a multi-item measure of self-reported urges to drink alcohol, predictor of drinking abuse and relapse. AUQ is an 8-item questionnaire.
  Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. Total score ranges from 8 to 56, and a higher score reflects greater craving.
Time Frame: 24 hours
Population: Data for this outcome measure were not collected for 1 participant in the ketamine arm and one participant in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Ketamine | Placebo
Number analyzed (Participants) | 16 | 10
score on a scale | 13.8 (12.2) | 16.3 (11.2)

5. Secondary Outcome: Manic Symptoms as Assessed by Score on the Young Mania Rating Scale (YMRS)
Description: The YMRS has 11 items, and total score ranges from 0 to 88, with a higher score indicating greater mania.
Time Frame: 24 hours
Population: Data for this outcome measure were not collected for 1 participant in the placebo arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Ketamine | Placebo
Number analyzed (Participants) | 17 | 10
score on a scale | 2.29 (2.85) | 2.40 (2.12)

6. Secondary Outcome: Dissociative State as Assessed by Score on Clinician-Administered Dissociative States Scale (CADSS)
Description: The CADSS consists of 23 items, and each item is rated on a scale from 0 (not at all) to 4 (severe), with the total score ranging from 0 to 92. A higher score indicates greater severity of dissociative state.
Time Frame: 24 hours
Population: Data for this outcome measure were not collected for 1 participant in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Ketamine | Placebo
Number analyzed (Participants) | 17 | 10
score on a scale | 0.824 (2.90) | 1.60 (3.20)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Intranasal Ketamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/11
Other Adverse Events (participants affected / at risk) | 12/17 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Ketamine (N=17) | Placebo (N=11)
Cognitive side effect (Nervous system disorders) | 12 (12) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03539887/Prot_SAP_000.pdf